CLINICAL TRIAL: NCT03766776
Title: Anlotinib Hydrochloride Capsules in the Treatment of Advanced Hepatocellular Carcinoma (HCC) Open, Single Arm, Exploratory Clinical Trial.
Brief Title: Anlotinib in the Treatment of Advanced Hepatocellular Carcinoma (HCC)
Acronym: ATAHC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-SR-273
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Cancer of Liver
MeSH Terms: conditions — Liver Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Arm (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib capsules: dosage of 12 mg PO qd, 14 days, 7 days, 21 days for a cycle. The dosage was adjusted according to the adverse reactions of patients.

SUMMARY:
This is a prospective, one-arm, exploratory clinical study to observe and evaluate the efficacy and safety of Anlotinib hydrochloride capsules in patients with advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years old.
* At least one measurable lesion (the length of spiral CT scan (> 10mm) meets the requirements of RESCIST 1.1) is found in patients with HCC confirmed by histopathology or cytology or who meet the clinical diagnostic criteria.
* Inability or unwillingness to undergo surgery and transcatheter hepatic artery interventional therapy; if interventional therapy, radiotherapy or surgery has been accepted, it must be more than 4 weeks, and adverse reactions or wounds have fully recovered.
* No treatment with sorafenib or other systemic treatment was received. Patients who have used interventional chemotherapeutic drugs during interventional therapy may be enrolled in the group.
* Child-Pugh liver function rating: grade A or B; BCLC stage B or C.
* ECOG PS：0-2.
* The life expectancy is more than 12 weeks.
* The main organs are functioning normally, which meets the following criteria:

  (1) Blood routine examination: A. HB > 90 g/L; (No blood transfusion within 14 days) B. ANC is more than 1.5 x /L; C. PLT is more than 50 x /L; (2) Biochemical examination: A. ALT and AST < 5_ULN; B. TBIL < 1.5_ULN; C. Plasma Cr < 1.5_ULN.
* Subjects volunteered to join the study, signed informed consent, good compliance, with follow-up.

Exclusion Criteria:

* Hepatobiliary and mixed cell carcinomas and fiberboard cell carcinomas are known; other malignant tumors (except cured cutaneous basal cell carcinomas and cervical carcinoma in situ) have been reported in the past or at the same time.
* Pregnant or lactating women .
* Patients with hypertension who could not be well controlled by antihypertensive drugs (systolic blood pressure > 150 mmHg, diastolic blood pressure > 100 mmHg), patients with myocardial ischemia or myocardial infarction above grade II, arrhythmias with poor control (including QTC interval > 450 ms) and cardiac insufficiency of grade III-IV according to NYHA standard.
* Inability to swallow, chronic diarrhea and intestinal obstruction significantly affect drug use and absorption.
* There are clear concerns about gastrointestinal bleeding (such as local active ulcer lesions, fecal occult blood +) or more), and there is a history of gastrointestinal bleeding within 6 months.
* Central nervous system metastasis has occurred.
* Coagulation dysfunction (PT > 16 s, APTT > 43 s, TT > 21 s, Fbg < 2 g/L), with bleeding tendency or undergoing thrombolysis or anticoagulation therapy.
* Have a history of mental illness or psychotropic drug abuse.
* Peritoneal effusion with clinical symptoms requires therapeutic abdominal puncture or drainage, or Child-Pugh score (> 2).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12-31 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 month
  Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongqian Shu, PhD, Study Chair — JANGSU PROVINCE HOSPITAL

IPD SHARING:
Plan to Share IPD: Undecided